CLINICAL TRIAL: NCT05753592
Title: A Phase 1, Open-label, Study to Investigate the Pharmacokinetics and Safety of Remibrutinib (LOU064) in Participants With Hepatic Impairment Compared to Matched Healthy Participants With Normal Hepatic Function
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Remibrutinib in Participants With Hepatic Impairment Compared With Matched Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064A2101; 2022-001936-27 (EudraCT Number)
Record Dates: First submitted 2022-10-11; First posted 2023-03-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Impairment
Keywords: Remibrutinib (LOU064); Hepatic Impairment (HI); Pharmacokinetic (PK); Safety; Tolerability; Child-Pugh
MeSH Terms: interventions — remibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1; LOU064 (Remibrutinib) (Experimental): Mild and Moderate HI participants and matching healthy participants
  Interventions: Drug: Part 1; LOU064 (Remibrutinib)
- Part 2; LOU064 (Remibrutinib) (Experimental): Severe HI participants and matching healthy participants
  Interventions: Drug: Part 2; LOU064 (Remibrutinib)

INTERVENTIONS:
Drug: Part 1; LOU064 (Remibrutinib) — 25 mg remibrutinib (5.5 days)
  Arms: Part 1; LOU064 (Remibrutinib)
Drug: Part 2; LOU064 (Remibrutinib) — 25 mg remibrutinib (5.5 days)
  Arms: Part 2; LOU064 (Remibrutinib)

SUMMARY:
This was a Phase 1, open-label study to evaluate the PK, safety, and tolerability after administration of multiple doses of remibrutinib in participants with mild, moderate, or severe hepatic impairment (HI) compared to pooled matched healthy control participants with normal hepatic function.

DETAILED DESCRIPTION:
This study was conducted in 2 parts. Part 1 was comprised of participants with mild (Child Pugh A; Group 1) and moderate (Child-Pugh B; Group 2) HI and matched healthy control participants with normal hepatic function (Group 4). Groups 1 and 2 were enrolled in parallel. Part 2 was comprised of participants with severe HI (Child-Pugh C; Group 3) and matched healthy control participants with normal hepatic function (Group 4). Matched healthy control participants (Group 4) were enrolled in parallel to Parts 1 and 2.

Up to 48 male and female participants, aged 18 to 70 years inclusive, were planned to be enrolled, with 8 participants enrolled in each of the mild (Child-Pugh A; Group 1 in Part 1), moderate (Child Pugh B; Group 2 in Part 1), and severe (Child-Pugh C; Group 3 in Part 2) HI groups, and up to 24 participants planned to be enrolled in the matched healthy control group (Group 4 from Parts 1 and 2). Additional participant(s) may have been enrolled if a participant discontinued from the study before completion of the PK assessment to ensure that at least 6 participants in each group completed the scheduled PK assessments. Due to difficulties in enrolling severe HI participants, only 7 severe HI participants were enrolled in this study.

Each study part was comprised of a screening period of up to 28 days (Day -29 to Day -2), a Baseline evaluation on Day -1, and a treatment period including up to 8 days of safety and PK data collection. Participants who met the eligibility criteria at Screening were admitted for Baseline evaluations on Day 1. Baseline safety assessments were performed prior to first dosing of study treatment. Participants were domiciled from Day -1 through Day 8.

All participants received 25 mg remibrutinib b.i.d. orally under fasting conditions on Days 1 and 2, and a morning oral dose of 25 mg remibrutinib on Day 3. PK samples were collected predose on Day 3 and until 72 hours post Day 3 dosing. Throughout the study, safety assessments included physical examinations, electrocardiograms (ECGs), vital signs, clinical laboratory evaluations (hematology, chemistry, urinalysis, and coagulation), and AE/serious adverse event (SAE) monitoring.

The investigator and Novartis conducted a joint interim review of safety and PK data from Part 1 before proceeding to Part 2. Data from at least 4 participants with mild HI (Group 1), 4 participants with moderate HI (Group 2), and their matched healthy control participants (Group 4), who completed PK study assessments up to Day 6 in Part 1, were evaluated.

Part 2 only began after administration of remibrutinib in the 4 evaluable participants from each of the mild and moderate HI groups (Groups 1 and 2) and their matched healthy control participants (Group 4) in Part 1 was deemed safe and tolerable based on the interim review by the investigator and Novartis. Depending on the outcome of the interim review, administration of a lower dose of remibrutinib in severe HI participants (Group 3) and their matched healthy control participants was to be considered. However, upon review of the interim data, the decision was made to not change the dose for severe HI participants.

As per the current study protocol, study drug strengths available for this trial were 25 mg and 10 mg. Therefore, the lowest dose that could have been used in Part 2 was 10 mg b.i.d. At the time of the interim data review, a decision was to be made as to whether or not to reduce the Part 2 dose, based on observed PK exposures and safety assessments in Part 1 and predicted exposures in severe HI participants in Part 2. In this particular case, Part 2 was to be initiated after the submission and approval of a Substantial Amendment from the respective Health Authorities (HA) and Ethics Committee (EC) were obtained. A decision was made to proceed with Part 2 using the same 25 mg dose as in Part 1.

Study Completion evaluations occurred on Day 8, followed by a post-study safety follow-up contact (e.g., follow-up telephone call, e-mail) approximately 30 days after last administration of study treatment. The information collected during the follow-up contact was kept as source documentation. The study was considered completed once all the participants finished the required assessments.

The total study duration for each participant was expected to be up to approximately 62 days, including the Screening period and the follow-up contact.

ELIGIBILITY:
Inclusion Criteria:

All participants

1. Signed informed consent was obtained prior to participation in the study.
2. Male and non-childbearing potential female* participants 18 to 70 years of age, inclusive, at Screening.
3. Women of non-childbearing potential were defined as women who were post menopausal or had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks prior to first dosing of study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman was confirmed by follow-up hormone level assessment was she considered not of childbearing potential. Women were considered post-menopausal if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms).
4. Must have been a non-smoker or a light smoker who smoked no more than 10 cigarettes (or equivalent) per day, at Screening. Smokers must have agreed to smoke no more than 5 cigarettes (or equivalent) per day from check-in until after Study Completion evaluations.
5. Must have been able to communicate well with the investigator and to understand and comply with the requirements of the study.

   Participants with mild, moderate, and severe HI (Groups 1, 2 and 3)
6. Must have weighed at least 50 kg to participate in the study and must have had a body mass index (BMI) within the range of 18.0 to 35.0 kg/m2, inclusive, at Screening.
7. Seated vital signs must have been within the following ranges at Screening and Baseline:

   * body temperature, 35.0 to 37.5°C, inclusive
   * systolic blood pressure (BP), 90 to 160 mmHg, inclusive
   * diastolic BP, 50 to 100 mmHg, inclusive
   * pulse rate, 50 to 110 bpm, inclusive
8. Had impaired hepatic function as defined by the Child-Pugh classification for severity of liver disease and had a Child-Pugh score in line with one of the following HI groups at Screening:

   * Group 1; mild (Class A); Child-Pugh score 5-6, inclusive
   * Group 2; moderate (Class B); Child-Pugh score 7-9, inclusive
   * Group 3; severe (Class C); Child-Pugh score 10-15, inclusive
9. Stable Child-Pugh status and no worsening of more than 1 point in Child-Pugh score within 28 days prior to first dosing of study treatment.
10. Participants with other stable medical disorders such as controlled diabetes, hyperlipidemia, hypothyroidism, etc., may have been eligible as long as they were considered appropriate for enrollment as determined by the investigator by past medical history, physical examination, ECG, and clinical laboratory tests at Screening.

    Healthy control participants (Group 4)
11. Each healthy participant must have matched the age (±10 years), body weight (±20%), and gender of at least one participant of Group 1 (Part 1), 2 (Part 1), or 3 (Part 2).
12. Must have weighed at least 50 kg to participate in the study and must have had a BMI within the range of 18.0 to 30.0 kg/m2, inclusive, at Screening.
13. Must have been in good health as determined by medical history, physical examination, ECG, and clinical laboratory tests at Screening.
14. Seated vital signs must have been within the following ranges at Screening and Baseline:

    * body temperature, 35.0 to 37.5°C, inclusive
    * systolic BP, 89 to 139 mmHg, inclusive
    * diastolic BP, 50 to 89 mmHg, inclusive
    * pulse rate, 45 to 90 bpm, inclusive

Exclusion Criteria:

All participants

1. Use of other investigational drugs within 5 half-lives or 30 days prior to first dosing of study treatment, whichever was longer.
2. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.
3. History or presence of malignancy of any organ system (other than treated localized basal cell or squamous cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years of Screening, regardless of whether there was evidence of local recurrence or metastases.
4. History of immunodeficiency diseases or had a positive human immunodeficiency virus (HIV) test result at Screening.
5. History or presence of any ongoing, chronic, or recurrent infectious disease (including tuberculosis, atypical mycobacterioses, listeriosis, aspergillosis).
6. Female participants who were of childbearing potential, defined as all women physiologically capable of becoming pregnant.
7. Female participants who were pregnant or nursing (lactating). Pregnancy was defined as the state of a female participant after conception and until termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test at Screening or Baseline.
8. Use of prohibited prescription or non-prescription medication or supplement.
9. Received any live vaccine within 8 weeks prior to first dosing of study treatment.
10. Received any coronavirus disease-2019 (COVID-19) vaccines within 2 weeks prior to first dosing of study treatment.
11. Clinical signs and symptoms consistent with COVID-19 (e.g., fever, dry cough, dyspnea, sore throat, fatigue) or confirmed infection by appropriate laboratory test within 2 weeks prior to Screening or tested positive during the Screening period before study site check in.
12. History or presence of significant bleeding risk or any coagulation disorder.
13. Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing of study treatment, or longer if required by local regulation.
14. Any surgical or medical condition which could have significantly altered the absorption, distribution, metabolism or excretion of drugs (apart from cholecystectomy), or which could have jeopardized the participants in case of participation in the study.
15. History of unhealthy alcohol use within 12 months prior to first dosing of study treatment, or evidence of such abuse as indicated by the laboratory assays (i.e., positive alcohol test) conducted during Screening or Baseline. Note: Participants who did not agree to comply with abstinence from alcohol use from 48 hours prior to first dosing of study treatment until after Study Completion evaluations were excluded. Unhealthy alcohol use was defined as a history of, or current alcohol misuse/abuse, defined as > 21 drinks for males and > 14 drinks for females in the same week.
16. Positive drug test at Screening or Baseline, unless the positive drug screen was due to prescription drug use that was approved by the investigator and Novartis.
17. Regular use of caffeine or methyl xanthine-containing products exceeding 800 mg (~4 cups of coffee containing 200 mg caffeine per cup) per day.

    Participants with mild and moderate HI (Groups 1 and 2)
18. Abnormal clinical laboratory values for any of the following parameters at Screening or Baseline:

    * hemoglobin < 9 g/dL
    * platelet count < 30 × 109/L
    * white blood cell count < 2.5 × 109/L
    * absolute neutrophil count < 1.5 × 109/L
    * lymphocytes < 0.8 × 109/L
    * total bilirubin (TBL) > 8 mg/dL
    * serum amylase > 2 × upper limit of normal (ULN)
    * INR > 2.3
    * serum ammonia level > 200 μg/dL
    * corrected serum calcium < 8.6 or > 10.2 mg/dL
19. Severe complications of liver disease within the preceding 3 months of Screening.
20. Emergency room visit or hospitalization due to liver disease within the preceding 3 months of Screening.
21. Received liver transplant at any time in the past and/or was on immunosuppressant therapy at Screening.
22. Required paracentesis more than every 30 days for the management of ascites.
23. Transjugular intrahepatic portosystemic shunt and/or underwent portacaval shunting.
24. Acute hepatitis B virus (HBV) or acute hepatitis C virus (HCV) infection. A positive hepatitis B surface antigen (HBsAg) test excluded a participant. Participants with a positive HCV antibody test had HCV ribonucleic acid (RNA) levels measured. Participants with positive (detectable) HCV RNA were excluded.
25. Clinically significant abnormal findings in physical examination, ECG or clinical laboratory evaluations, not consistent with known liver disease. Participants having had myocardial infarction < 5 years of Screening were not eligible to participate; participants having had myocardial infarction ≥ 5 years of Screening could have been eligible to participate.
26. Presence of moderate to severe impaired renal function as indicated by any of the following at Screening:

    * Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
    * Serum creatinine > 1.5 × ULN
27. Encephalopathy Grade 3 or worse within 28 days of planned first dosing of study treatment.
28. Primary biliary cholangitis or biliary obstruction.
29. History of gastrointestinal (GI) bleeding within the past 3 months prior to Screening.
30. Clinically significant illness within 2 weeks prior to first dosing that could have jeopardized safety of the study participant and/or altered the study results as judged by the investigator.

    Participants with severe HI (Group 3)
31. Abnormal clinical laboratory values for any of the following parameters at Screening or Baseline:

    * hemoglobin < 8.5 g/dL
    * platelet count < 30 × 109/L
    * white blood cell count < 2.5 × 109/L
    * TBL > 8 mg/dL
    * serum amylase > 2 × ULN
    * serum ammonia level > 200 μg/dL
    * INR > 2.3
32. Severe complications of liver disease within the preceding 3 months of Screening.
33. Emergency room visit or hospitalization due to liver disease within the preceding 1 month of Screening.
34. Received liver transplant at any time in the past and/or was on immunosuppressant therapy at Screening.
35. Required paracentesis more than every 30 days for the management of ascites.
36. Transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.
37. Acute HBV or acute HCV infection. A positive HBsAg test excluded a participant. Participants with a positive HCV antibody test had HCV RNA levels measured. Participants with positive (detectable) HCV RNA were excluded.
38. Clinically significant abnormal findings in physical examination, ECG or clinical laboratory evaluations, not consistent with known liver disease. Participants having had myocardial infarction < 5 years of Screening were not eligible to participate, participants having had myocardial infarction ≥ 5 years of Screening could have been eligible to participate.
39. Presence of moderate to severe impaired renal function as indicated by any of the following at Screening:

    * eGFR < 45 mL/min/1.73 m2 based on the CKD-EPI equation
    * Serum creatinine > 1.5 × ULN
40. Encephalopathy Grade 3 or worse within 28 days of planned first dosing of study treatment.
41. Primary biliary cholangitis or biliary obstruction.
42. History of GI bleeding within the past 3 months prior to Screening.
43. Documented presence of esophageal varices (Stage 3 or 4) based on the evaluation of the participant's medical history at Screening and Baseline.
44. History, clinical evidence or suspicion of a hepato-cellular carcinoma (HCC) based on sonographical and/or laboratory results (i.e., α-fetoprotein [AFP] > 12 IU/mL [2 × ULN] at Screening).
45. Severe ascites and/or pleural effusion.
46. Participants with clinical evidence of suspected acute liver failure as judged by the investigator.
47. Clinically significant illness within 2 weeks prior to first dosing that could have jeopardized safety of the study participant and/or altered the study results as judged by the investigator.

    Healthy control participants (Group 4)
48. Significant illness which had not resolved within 2 weeks prior to first dosing of study treatment.
49. Liver disease or liver injury as indicated by abnormal liver function tests at Screening. Any single parameter of alanine aminotransferase (ALT), AST, gamma-glutamyltransferase (GGT), or alkaline phosphatase (ALP) exceeding 1.2 × ULN or ≥ 1.5 × ULN TBL OR any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP or TBL.
50. Known to have Gilbert's syndrome.
51. Positive result for HBsAg or HCV antibody at Screening.
52. Hemoglobin levels below 11.0 g/dL for males and 10.0 g/dL for females at Screening or Baseline.
53. History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or blood urea nitrogen (BUN) and/or urea values, or abnormal urinary constituents at Screening.

In the case where a safety laboratory assessment at Screening or Baseline was outside of the range specified above, the assessment may have been repeated once at Screening and/or once at Baseline. If the repeat value remained outside of the specified ranges, the participant was excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | 72 hours
  The maximum (peak) observed blood concentration following multiple-dose administration (mass/volume)
AUCtau | 72 hours
  The area under the curve (AUC) from time zero to the end of the dosing interval tau (12 hours) following multiple-dose administration
AUClast,ss | 72 hours
  The area under the curve (AUC) from time zero to the last measurable blood concentration sampling time (Tlast) following multiple-dose administration (mass*time/volume)
Tmax,ss | 72 hours
  The time to reach maximum (peak) blood concentration following multiple-dose administration (time)
T1/2 | 72 hours
  The elimination half-life associated with the terminal slope (lambda_z) of a semi logarithmic concentration-time curve (time)

SECONDARY OUTCOMES:
Number of participants with adverse events | 8 days
  The distribution of adverse events was done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Unbound fraction; Cmax,ss,u | 8 days
  The maximum (peak) observed unbound plasma concentration following multiple-dose administration (mass/volume)
Unbound fraction; AUCtau,u | 8 days
  The unbound plasma AUC from time zero to the end of the dosing interval tau (12 hours) following multiple-dose administration
Unbound fraction; AUClast,ss,u | 8 days
  The area under the curve (AUC) from time zero to the last measurable unbound plasma concentration sampling time (Tlast) following multiple-dose administration (mass*time/volume)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Miskolc, Baz, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2414